CLINICAL TRIAL: NCT01440621
Title: Randomized Controlled Study to Evaluate the Effects of Modafinil in Cancer Related Fatigue in Patients Undergoing Radiation Therapy
Brief Title: Modafinil in Cancer Related Fatigue
Acronym: ModCRF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indira Gandhi Medical College, Shimla (Other)
Responsible Party: Principal Investigator, Swaroop Revannasiddaiah, Post-Graduate in Radiation Oncology, Indira Gandhi Medical College, Shimla
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ModCRF
Record Dates: First submitted 2011-09-20; First posted 2011-09-26 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Cancer Related Fatigue; Quality of Life
Keywords: Cancer related fatigue; Quality of life; Modafinil; Radiation therapy; Radiotherapy
MeSH Terms: interventions — Modafinil; Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Arm M (Active Comparator): Will be treated with Tab Modafinil (generic) 100mg Once a Day in the Morning starting from Day 1 of RT till the first follow-up.
  Interventions: Drug: Modafinil
- Arm P (Placebo Comparator): Will be given placebo (Tab Pyridoxine 10mg) which physically resembles Tab Modafinil 100mg.
  Interventions: Drug: Pyridoxine

INTERVENTIONS:
Drug: Modafinil — Tablet Modafinil 100mg (Generic) to be given in 100mg once a day dose, at 8AM daily in the morning, and to be given from Day 1 of Radiation Therapy till the first post treatment follow-up
  Arms: Arm M
Drug: Pyridoxine — Tablet Pyridoxine 10mg once a day at 8AM daily, from Day one of RT till first post-treatment followup. Tab Pyridoxine 10mg has been chosen as placebo as it resembles Tab Modafinil 100mg in physical appearance, size and shape. Tab Pyridoxine is unlikely to affect Cancer Related Fatigue on its own as all patients on RT are already on multivitamin supplements as per our institutional guidelines.
  Arms: Arm P

SUMMARY:
Cancer related fatigue (CRF) is a highly prevalent and highly significant entity among patients with cancer. 'Cancer related fatigue' is not a simple symptom, but is an entity in itself, in that it is different from routine fatigue. Cancer related fatigue is that fatigue which persists even after rest and has significant effects on quality of life.

The incidence of Cancer Related Fatigue (CRF) increases during radiation therapy (RT), with almost every patient on radiotherapy complaining of at-least some magnitude of fatigue.

Given that fatigue can affect treatment adherence by patients, it is important to initiate measures to either prevent or mitigate Cancer Related Fatigue.

The investigators intend to use modafinil in cancer related fatigue, in view of the fact that it has safety and efficacy in other diseases such as narcolepsy, multiple sclerosis and fibromyalgia. In addition, there have been a few small trials which have hinted towards benefit with the use of modafinil in cancer related fatigue.

The investigators have chosen a dose of 100mg/day in the morning, to be compared with placebo. The study arm and the placebo arm will be stratified with respect to age, sex, disease site, baseline performance status.

Primary outcome would be fatigue, which will be assessed by the use of Brief Fatigue Inventory (BFI). Secondary outcomes include Quality of Life, improvements in performance status, changes in systolic and diastolic blood pressure, and changes in weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological confirmation of cancer
* Age 18 years to 70 years
* Performance status (Karnofsky scale) not less than 60
* Providing consent

Exclusion Criteria:

* Psychiatric illness
* Hypertension
* Diabetes
* Thyroid disorders
* Epilepsy
* Tuberculosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction in Cancer Related Fatigue | Baseline and 12 weeks
  Changes in Fatigue measured with the Brief Fatigue Inventory (BFI).

SECONDARY OUTCOMES:
Improvement in Quality of Life | Baseline and 12 weeks
  The Spitzer Quality of Life Index (SQLI) to obtain Quality of Life (QOL) measurements.
Karnofsky Performance Status Scores | Baseline and 12 weeks
  Performance status scores measured with the Karnofsky Performance Status (KPS) scale.
Effects of Modafinil on Systolic and Diastolic Blood Pressure | Baseline and 12 weeks
Changes in weight | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Cancer Centre, Shimla, Himachal Pradesh, India

REFERENCES:
- [Result] Spathis A, Dhillan R, Booden D, Forbes K, Vrotsou K, Fife K. Modafinil for the treatment of fatigue in lung cancer: a pilot study. Palliat Med. 2009 Jun;23(4):325-31. doi: 10.1177/0269216309102614. Epub 2009 Mar 6. PMID 19270033
- [Result] Cooper MR, Bird HM, Steinberg M. Efficacy and safety of modafinil in the treatment of cancer-related fatigue. Ann Pharmacother. 2009 Apr;43(4):721-5. doi: 10.1345/aph.1L532. Epub 2009 Mar 24. PMID 19318599
- [Result] Blackhall L, Petroni G, Shu J, Baum L, Farace E. A pilot study evaluating the safety and efficacy of modafinal for cancer-related fatigue. J Palliat Med. 2009 May;12(5):433-9. doi: 10.1089/jpm.2008.0230. PMID 19416039
- [Result] Wirz S, Nadstawek J, Kuhn KU, Vater S, Junker U, Wartenberg HC. [Modafinil for the treatment of cancer-related fatigue : an intervention study]. Schmerz. 2010 Dec;24(6):587-95. doi: 10.1007/s00482-010-0987-y. German. PMID 21046171
- [Result] Jean-Pierre P, Morrow GR, Roscoe JA, Heckler C, Mohile S, Janelsins M, Peppone L, Hemstad A, Esparaz BT, Hopkins JO. A phase 3 randomized, placebo-controlled, double-blind, clinical trial of the effect of modafinil on cancer-related fatigue among 631 patients receiving chemotherapy: a University of Rochester Cancer Center Community Clinical Oncology Program Research base study. Cancer. 2010 Jul 15;116(14):3513-20. doi: 10.1002/cncr.25083. PMID 20564068
- See also: Link to a trial which utilized modafinil as an intervention for cancer related fatigue in 631 patients of breast cancer undergoing chemo — http://www.ncbi.nlm.nih.gov/pubmed/20564068
- See also: A small study which showed that modafinil was well-tolerated and effective for fatigue in patients with cancer. — http://www.ncbi.nlm.nih.gov/pubmed/19416039
- See also: A study which called for randomized trials with modafinil in cancer related fatigue — http://www.ncbi.nlm.nih.gov/pubmed/19318599
- See also: Link to an article validating the Brief Fatigue Inventory (scale for fatigue assessment). — http://www.ncbi.nlm.nih.gov/pubmed/10091805